CLINICAL TRIAL: NCT01315639
Title: Plasma Abeta Peptides and the Risk of Alzheimer's Disease. Diagnostic Performance and Predictive and Prognostic Values of Measurements of Plasma Amyloid Peptides Concentrations for the Diagnosis of Alzheimer's Disease
Brief Title: New Biomarker for Alzheimer's Disease Diagnostic
Acronym: BALTAZAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P081205
Record Dates: First submitted 2011-03-11; First posted 2011-03-15 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
Keywords: Dementia; Cognitive impairment; Memory impairment; Mild Cognitive Impairment; Cerebrospinal fluid; Plasma; Biomarker; Longitudinal; Abeta peptide amyloid, saPP alpha; Oculomotor impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia; Memory Disorders | interventions — Biomarkers; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- biomarkers, MRI and CSF (Other): Longitudinal multicenter study including 1300 subjects with amnestic impairment (MCI, n=650 and AD, n=650) derived from the main French national Memory Resources and Research Centers.
  Participants will undergo at baseline and every 6 months a neurological examination, a neuropsychological assessment (and an oculomotor examination for those included from Broca Hospital).
  Alzheimer disease biomarkers' measurements will be performed at inclusion and at the end of the study (or the conversion).
  Interventions: Biological: biomarkers, MRI and CSF

INTERVENTIONS:
Biological: biomarkers, MRI and CSF — MRI at Day 0 and month 24 (or conversion) Biomarkers at Day 0 et month 24 (or conversion) CSF at D0

SUMMARY:
The aim of this study is to examine the relationship between plasma putative biomarkers for Alzheimer's disease (i.e. Ab40 amyloid and total Ab42 amyloid, free, bound, free/bound, truncated, sAPPα) and :

* the risk of conversion of individuals with Mild Cognitive Impairment (MCI) into Alzheimer's disease (AD),
* the Alzheimer's disease progression rate.

DETAILED DESCRIPTION:
Rational Whether there are biological markers of Alzheimer's disease (AD) is crucial for adequate targeting and appropriate management of the disease. The aim of our study is to examine diagnostic performance and predictive and prognostic values of new plasma markers of AD.

Results of studies on the predictive value of plasma concentrations of Aβ40 and 42 amyloid peptides for incident AD are not straightforward. Discrepancies in these results may be due to the fact that total peptide concentrations have been measured. One recent study suggests that plasma free Aβ peptide concentration and particularly low-density lipoprotein receptor-related protein (LPR) as like as free Aβ/total Aβ ratio would be more reliable and discriminant.

Main objective of the study To examine the association between plasma free Aβ peptide concentration and (1) the risk of conversion of subjects with Mild Cognitive Impairment (MCI) into Alzheimer's disease (AD) and (2) the risk of worsening of the disease in patients with mild and moderate stages of AD.

Secondary objectives

* To examine the association of total peptid Aβ concentration, free Aβ/Total Aβ ratio, and trunked plasmatic Aβ to the risk of incident AD in MCI subjects, and to the risk of worsening of the disease in mild and moderate AD patients,
* To examine the association between serum sAPP concentration and the risk of incident AD in MCI subjects, and the risk of worsening of the disease in mild and moderate AD patients,
* To compare the time evolution of concentrations of these biomarkers to Alzheimer's disease progression rate which will be assessed on the basis of neuropsychological examinations and MRI examination of hippocampal atrophy,
* To examine the association between serum and cerebrospinal fluid (CSF) concentrations of AD biomarkers in subgroup of participants who undergo lumbar puncture,
* To examine the association between neuroimaging data (cerebral volume, hippocampal volume, cerebrovascular lesions and plasma and CSF AD biomarkers' concentrations,
* To constitute blood and plasma banks, gene bank and CSF bank for future studies on other biomarkers of AD.

Design and Methods Longitudinal multicenter study including 1300 subjects with amnestic impairment (MCI, n=650 and AD, n=650) derived from the main French national Memory Resources and Research Centers.

Participants will undergo at baseline and every 6 months a neurological examination, a neuropsychological assessment (and an oculomotor examination for those included from Broca Hospital).

Alzheimer disease biomarkers' measurements will be performed at inclusion and at the end of the study. For those MCI participants who convert to dementia, the end of the study will correspond to the AD conversion period.

A Magnetic Resonance Imaging (MRI) scan will be performed at inclusion and at the end of the study for MCI subjects who convert into AD.

A lumbar puncture on an outpatient basis will be performed at study entry in all participants who will give an informed consent for this examination in absence of contraindication.

ELIGIBILITY:
Inclusion Criteria:

MCI group :

* ≥ 70 years
* MCI diagnosis : New criteria (Petersen, PORTET*)

  1. cognitive complaint from the patient, family, or both,
  2. report by the subject or reporter of a decline in cognitive or functional performance, relative to previous abilities,
  3. cognitive disorders evidenced by clinical evaluation: impairment in memory or another cognitive domain,
  4. cognitive impairment without any repercussion on daily life, even if the subject reports difficulties concerning complex daily activities,
  5. no dementia
* Having signed an informed consent form
* Fluent in French

AD group :

* ≥ 45 years
* AD diagnosis (DSM IV-TR et NINCDS-ADRDA)
* Mild to moderate (MMSE > 15)
* Having signed an informed consent form
* Caregiver/informant to provide information on patient

Exclusion Criteria:

* Normal cognitive function
* Major depression (according to the DSMIV-TR or MINI or Geriatric depression Scale> 20/30)
* Genetic form of AD (genetic mutation known)
* All other diseases that could interfere with cognitive assessment (Epilepsy, Parkinson's disease, schizophrenia, other dementia)
* Major sensory deficits that could interfere with cognitive assessment (visual and auditory)
* Diseases involving the short-term survival (advanced cancer, unstable heart disease, severe hepatic/respiratory/renal failure)
* Contraindication for MRI, for lumbar puncture (i.e. anticoagulant agents)
* Use of any experimental agent for the duration of the study
* Participation to other biomedical research that could interfere with principal objective of the study
* For MCI patient, use of IchE or memantine medication before inclusion
* Less than 4 years of education
* Illiteracy, is unable to count or to read
* Pregnant women
* Non health insurance affiliation
* Private subjects of freedom by legal or administrative decision
* Contraindication for MRI examination:
* Claustrophobic subject
* Carrying a cardiac pacemaker
* Presence of any ferromagnetic metallic implants or foreign bodies (carrying an internal electrical/magnetic device, carrying a valvular prosthesis)
* Carrying a ventricular valvular

Exclusion criteria specific to the lumbar puncture:

• Taking anticoagulant agents

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1067 (Actual)
Dates: Start 2010-09-03 (Actual); Primary Completion 2015-02-26 (Actual); Study Completion 2018-03-16 (Actual)

PRIMARY OUTCOMES:
Mean concentration of plasma AB peptides | at t0 and 24 months
  * MCI "converted" (MCI-AD)
  * and stable MCI (MCI-MCI) groups
plasma levels of Tau protein | t0
  Ancillary study :comparison of plasma levels of Tau protein at baseline between MCI converters and MCI non-converters and between rapidly and non-rapidly progressing AD.

SECONDARY OUTCOMES:
Mean concentration of biomarker | t0 and 24 months
  * Mean plasma concentration of AB peptides between
    * fast decliner AD (decline of 7 points or more in ADAS-cog)
    * and non fast decliner AD groups
  * Mean concentration of sAPPalpha between
    * MCI "converted" (MCI-AD)
    * and stable MCI (MCI-MCI) groups
  * Mean concentration of sAPPalpha between
    * fast decliner AD (decline of 7 points or more in ADAS-cog)
    * and non fast decliner AD groups
MRI | T0 + M24 or conversion
  •Relationship between MRI measures (brain volume, hippocampus atrophy, vascular lesions) and biomarkers
Transcriptomics biomarkers | T0 and 24 months or conversions
  • Relationship between transcriptomics biomarkers and cognitive decline
Bace peptide | t0
  ancillary study
TACE/ADAM17 | to
  ancillary study
Cathepsin | t0
  ancillary study
sAPPβ | t0
  ancillary study
Ratio of CSF sAPPβ and CSF sAPPα | t0
  ancillary study
Ratio of plasma Aβ and plasma Tau | t0
  ancillary study
Plasma Tau | 24 months
  ancillary study
MRI biomarkers | t0
  ancillary study
MRI biomarkers | 24 months
  ancillary study

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Hanon, ph, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- APHP, Hôpital Broca, Paris, France

REFERENCES:
- [Background] Hanon O, Vidal JS, Lehmann S, Bombois S, Allinquant B, Treluyer JM, Gele P, Delmaire C, Blanc F, Mangin JF, Buee L, Touchon J, Hugon J, Vellas B, Galbrun E, Benetos A, Berrut G, Paillaud E, Wallon D, Castelnovo G, Volpe-Gillot L, Paccalin M, Robert PH, Godefroy O, Dantoine T, Camus V, Belmin J, Vandel P, Novella JL, Duron E, Rigaud AS, Schraen-Maschke S, Gabelle A; BALTAZAR study group. Plasma amyloid levels within the Alzheimer's process and correlations with central biomarkers. Alzheimers Dement. 2018 Jul;14(7):858-868. doi: 10.1016/j.jalz.2018.01.004. Epub 2018 Feb 17. PMID 29458036
- [Background] Hanon O, Vidal JS, Lehmann S, Bombois S, Allinquant B, Baret-Rose C, Treluyer JM, Abdoul H, Gele P, Delmaire C, Blanc F, Mangin JF, Buee L, Touchon J, Hugon J, Vellas B, Galbrun E, Benetos A, Berrut G, Paillaud E, Wallon D, Castelnovo G, Volpe-Gillot L, Paccalin M, Robert P, Godefroy O, Camus V, Belmin J, Vandel P, Novella JL, Duron E, Rigaud AS, Schraen-Maschke S, Gabelle A; BALTAZAR study group. Plasma amyloid beta predicts conversion to dementia in subjects with mild cognitive impairment: The BALTAZAR study. Alzheimers Dement. 2022 Dec;18(12):2537-2550. doi: 10.1002/alz.12613. Epub 2022 Feb 20. PMID 35187794
- [Background] Duron E, Vidal JS, Grousselle D, Gabelle A, Lehmann S, Pasquier F, Bombois S, Buee L, Allinquant B, Schraen-Maschke S, Baret C, Rigaud AS, Hanon O, Epelbaum J. Corrigendum: Somatostatin and Neuropeptide Y in Cerebrospinal Fluid: Correlations With Amyloid Peptides Ass1-42, and Tau Proteins in Elderly Patients With Mild Cognitive Impairment. Front Aging Neurosci. 2019 Feb 19;11:11. doi: 10.3389/fnagi.2019.00011. eCollection 2019. PMID 30837862
- [Background] Kunkle BW, Grenier-Boley B, Sims R, Bis JC, Damotte V, Naj AC, Boland A, Vronskaya M, van der Lee SJ, Amlie-Wolf A, Bellenguez C, Frizatti A, Chouraki V, Martin ER, Sleegers K, Badarinarayan N, Jakobsdottir J, Hamilton-Nelson KL, Moreno-Grau S, Olaso R, Raybould R, Chen Y, Kuzma AB, Hiltunen M, Morgan T, Ahmad S, Vardarajan BN, Epelbaum J, Hoffmann P, Boada M, Beecham GW, Garnier JG, Harold D, Fitzpatrick AL, Valladares O, Moutet ML, Gerrish A, Smith AV, Qu L, Bacq D, Denning N, Jian X, Zhao Y, Del Zompo M, Fox NC, Choi SH, Mateo I, Hughes JT, Adams HH, Malamon J, Sanchez-Garcia F, Patel Y, Brody JA, Dombroski BA, Naranjo MCD, Daniilidou M, Eiriksdottir G, Mukherjee S, Wallon D, Uphill J, Aspelund T, Cantwell LB, Garzia F, Galimberti D, Hofer E, Butkiewicz M, Fin B, Scarpini E, Sarnowski C, Bush WS, Meslage S, Kornhuber J, White CC, Song Y, Barber RC, Engelborghs S, Sordon S, Voijnovic D, Adams PM, Vandenberghe R, Mayhaus M, Cupples LA, Albert MS, De Deyn PP, Gu W, Himali JJ, Beekly D, Squassina A, Hartmann AM, Orellana A, Blacker D, Rodriguez-Rodriguez E, Lovestone S, Garcia ME, Doody RS, Munoz-Fernadez C, Sussams R, Lin H, Fairchild TJ, Benito YA, Holmes C, Karamujic-Comic H, Frosch MP, Thonberg H, Maier W, Roshchupkin G, Ghetti B, Giedraitis V, Kawalia A, Li S, Huebinger RM, Kilander L, Moebus S, Hernandez I, Kamboh MI, Brundin R, Turton J, Yang Q, Katz MJ, Concari L, Lord J, Beiser AS, Keene CD, Helisalmi S, Kloszewska I, Kukull WA, Koivisto AM, Lynch A, Tarraga L, Larson EB, Haapasalo A, Lawlor B, Mosley TH, Lipton RB, Solfrizzi V, Gill M, Longstreth WT Jr, Montine TJ, Frisardi V, Diez-Fairen M, Rivadeneira F, Petersen RC, Deramecourt V, Alvarez I, Salani F, Ciaramella A, Boerwinkle E, Reiman EM, Fievet N, Rotter JI, Reisch JS, Hanon O, Cupidi C, Andre Uitterlinden AG, Royall DR, Dufouil C, Maletta RG, de Rojas I, Sano M, Brice A, Cecchetti R, George-Hyslop PS, Ritchie K, Tsolaki M, Tsuang DW, Dubois B, Craig D, Wu CK, Soininen H, Avramidou D, Albin RL, Fratiglioni L, Germanou A, Apostolova LG, Keller L, Koutroumani M, Arnold SE, Panza F, Gkatzima O, Asthana S, Hannequin D, Whitehead P, Atwood CS, Caffarra P, Hampel H, Quintela I, Carracedo A, Lannfelt L, Rubinsztein DC, Barnes LL, Pasquier F, Frolich L, Barral S, McGuinness B, Beach TG, Johnston JA, Becker JT, Passmore P, Bigio EH, Schott JM, Bird TD, Warren JD, Boeve BF, Lupton MK, Bowen JD, Proitsi P, Boxer A, Powell JF, Burke JR, Kauwe JSK, Burns JM, Mancuso M, Buxbaum JD, Bonuccelli U, Cairns NJ, McQuillin A, Cao C, Livingston G, Carlson CS, Bass NJ, Carlsson CM, Hardy J, Carney RM, Bras J, Carrasquillo MM, Guerreiro R, Allen M, Chui HC, Fisher E, Masullo C, Crocco EA, DeCarli C, Bisceglio G, Dick M, Ma L, Duara R, Graff-Radford NR, Evans DA, Hodges A, Faber KM, Scherer M, Fallon KB, Riemenschneider M, Fardo DW, Heun R, Farlow MR, Kolsch H, Ferris S, Leber M, Foroud TM, Heuser I, Galasko DR, Giegling I, Gearing M, Hull M, Geschwind DH, Gilbert JR, Morris J, Green RC, Mayo K, Growdon JH, Feulner T, Hamilton RL, Harrell LE, Drichel D, Honig LS, Cushion TD, Huentelman MJ, Hollingworth P, Hulette CM, Hyman BT, Marshall R, Jarvik GP, Meggy A, Abner E, Menzies GE, Jin LW, Leonenko G, Real LM, Jun GR, Baldwin CT, Grozeva D, Karydas A, Russo G, Kaye JA, Kim R, Jessen F, Kowall NW, Vellas B, Kramer JH, Vardy E, LaFerla FM, Jockel KH, Lah JJ, Dichgans M, Leverenz JB, Mann D, Levey AI, Pickering-Brown S, Lieberman AP, Klopp N, Lunetta KL, Wichmann HE, Lyketsos CG, Morgan K, Marson DC, Brown K, Martiniuk F, Medway C, Mash DC, Nothen MM, Masliah E, Hooper NM, McCormick WC, Daniele A, McCurry SM, Bayer A, McDavid AN, Gallacher J, McKee AC, van den Bussche H, Mesulam M, Brayne C, Miller BL, Riedel-Heller S, Miller CA, Miller JW, Al-Chalabi A, Morris JC, Shaw CE, Myers AJ, Wiltfang J, O'Bryant S, Olichney JM, Alvarez V, Parisi JE, Singleton AB, Paulson HL, Collinge J, Perry WR, Mead S, Peskind E, Cribbs DH, Rossor M, Pierce A, Ryan NS, Poon WW, Nacmias B, Potter H, Sorbi S, Quinn JF, Sacchinelli E, Raj A, Spalletta G, Raskind M, Caltagirone C, Bossu P, Orfei MD, Reisberg B, Clarke R, Reitz C, Smith AD, Ringman JM, Warden D, Roberson ED, Wilcock G, Rogaeva E, Bruni AC, Rosen HJ, Gallo M, Rosenberg RN, Ben-Shlomo Y, Sager MA, Mecocci P, Saykin AJ, Pastor P, Cuccaro ML, Vance JM, Schneider JA, Schneider LS, Slifer S, Seeley WW, Smith AG, Sonnen JA, Spina S, Stern RA, Swerdlow RH, Tang M, Tanzi RE, Trojanowski JQ, Troncoso JC, Van Deerlin VM, Van Eldik LJ, Vinters HV, Vonsattel JP, Weintraub S, Welsh-Bohmer KA, Wilhelmsen KC, Williamson J, Wingo TS, Woltjer RL, Wright CB, Yu CE, Yu L, Saba Y, Pilotto A, Bullido MJ, Peters O, Crane PK, Bennett D, Bosco P, Coto E, Boccardi V, De Jager PL, Lleo A, Warner N, Lopez OL, Ingelsson M, Deloukas P, Cruchaga C, Graff C, Gwilliam R, Fornage M, Goate AM, Sanchez-Juan P, Kehoe PG, Amin N, Ertekin-Taner N, Berr C, Debette S, Love S, Launer LJ, Younkin SG, Dartigues JF, Corcoran C, Ikram MA, Dickson DW, Nicolas G, Campion D, Tschanz J, Schmidt H, Hakonarson H, Clarimon J, Munger R, Schmidt R, Farrer LA, Van Broeckhoven C, C O'Donovan M, DeStefano AL, Jones L, Haines JL, Deleuze JF, Owen MJ, Gudnason V, Mayeux R, Escott-Price V, Psaty BM, Ramirez A, Wang LS, Ruiz A, van Duijn CM, Holmans PA, Seshadri S, Williams J, Amouyel P, Schellenberg GD, Lambert JC, Pericak-Vance MA; Alzheimer Disease Genetics Consortium (ADGC),; European Alzheimer's Disease Initiative (EADI),; Cohorts for Heart and Aging Research in Genomic Epidemiology Consortium (CHARGE),; Genetic and Environmental Risk in AD/Defining Genetic, Polygenic and Environmental Risk for Alzheimer's Disease Consortium (GERAD/PERADES),. Genetic meta-analysis of diagnosed Alzheimer's disease identifies new risk loci and implicates Abeta, tau, immunity and lipid processing. Nat Genet. 2019 Mar;51(3):414-430. doi: 10.1038/s41588-019-0358-2. Epub 2019 Feb 28. PMID 30820047
- [Background] de Rojas I, Moreno-Grau S, Tesi N, Grenier-Boley B, Andrade V, Jansen IE, Pedersen NL, Stringa N, Zettergren A, Hernandez I, Montrreal L, Antunez C, Antonell A, Tankard RM, Bis JC, Sims R, Bellenguez C, Quintela I, Gonzalez-Perez A, Calero M, Franco-Macias E, Macias J, Blesa R, Cervera-Carles L, Menendez-Gonzalez M, Frank-Garcia A, Royo JL, Moreno F, Huerto Vilas R, Baquero M, Diez-Fairen M, Lage C, Garcia-Madrona S, Garcia-Gonzalez P, Alarcon-Martin E, Valero S, Sotolongo-Grau O, Ullgren A, Naj AC, Lemstra AW, Benaque A, Perez-Cordon A, Benussi A, Rabano A, Padovani A, Squassina A, de Mendonca A, Arias Pastor A, Kok AAL, Meggy A, Pastor AB, Espinosa A, Corma-Gomez A, Martin Montes A, Sanabria A, DeStefano AL, Schneider A, Haapasalo A, Kinhult Stahlbom A, Tybjaerg-Hansen A, Hartmann AM, Spottke A, Corbaton-Anchuelo A, Rongve A, Borroni B, Arosio B, Nacmias B, Nordestgaard BG, Kunkle BW, Charbonnier C, Abdelnour C, Masullo C, Martinez Rodriguez C, Munoz-Fernandez C, Dufouil C, Graff C, Ferreira CB, Chillotti C, Reynolds CA, Fenoglio C, Van Broeckhoven C, Clark C, Pisanu C, Satizabal CL, Holmes C, Buiza-Rueda D, Aarsland D, Rujescu D, Alcolea D, Galimberti D, Wallon D, Seripa D, Grunblatt E, Dardiotis E, Duzel E, Scarpini E, Conti E, Rubino E, Gelpi E, Rodriguez-Rodriguez E, Duron E, Boerwinkle E, Ferri E, Tagliavini F, Kucukali F, Pasquier F, Sanchez-Garcia F, Mangialasche F, Jessen F, Nicolas G, Selbaek G, Ortega G, Chene G, Hadjigeorgiou G, Rossi G, Spalletta G, Giaccone G, Grande G, Binetti G, Papenberg G, Hampel H, Bailly H, Zetterberg H, Soininen H, Karlsson IK, Alvarez I, Appollonio I, Giegling I, Skoog I, Saltvedt I, Rainero I, Rosas Allende I, Hort J, Diehl-Schmid J, Van Dongen J, Vidal JS, Lehtisalo J, Wiltfang J, Thomassen JQ, Kornhuber J, Haines JL, Vogelgsang J, Pineda JA, Fortea J, Popp J, Deckert J, Buerger K, Morgan K, Fliessbach K, Sleegers K, Molina-Porcel L, Kilander L, Weinhold L, Farrer LA, Wang LS, Kleineidam L, Farotti L, Parnetti L, Tremolizzo L, Hausner L, Benussi L, Froelich L, Ikram MA, Deniz-Naranjo MC, Tsolaki M, Rosende-Roca M, Lowenmark M, Hulsman M, Spallazzi M, Pericak-Vance MA, Esiri M, Bernal Sanchez-Arjona M, Dalmasso MC, Martinez-Larrad MT, Arcaro M, Nothen MM, Fernandez-Fuertes M, Dichgans M, Ingelsson M, Herrmann MJ, Scherer M, Vyhnalek M, Kosmidis MH, Yannakoulia M, Schmid M, Ewers M, Heneka MT, Wagner M, Scamosci M, Kivipelto M, Hiltunen M, Zulaica M, Alegret M, Fornage M, Roberto N, van Schoor NM, Seidu NM, Banaj N, Armstrong NJ, Scarmeas N, Scherbaum N, Goldhardt O, Hanon O, Peters O, Skrobot OA, Quenez O, Lerch O, Bossu P, Caffarra P, Dionigi Rossi P, Sakka P, Mecocci P, Hoffmann P, Holmans PA, Fischer P, Riederer P, Yang Q, Marshall R, Kalaria RN, Mayeux R, Vandenberghe R, Cecchetti R, Ghidoni R, Frikke-Schmidt R, Sorbi S, Hagg S, Engelborghs S, Helisalmi S, Botne Sando S, Kern S, Archetti S, Boschi S, Fostinelli S, Gil S, Mendoza S, Mead S, Ciccone S, Djurovic S, Heilmann-Heimbach S, Riedel-Heller S, Kuulasmaa T, Del Ser T, Lebouvier T, Polak T, Ngandu T, Grimmer T, Bessi V, Escott-Price V, Giedraitis V, Deramecourt V, Maier W, Jian X, Pijnenburg YAL; EADB contributors; GR@ACE study group; DEGESCO consortium; IGAP (ADGC, CHARGE, EADI, GERAD); PGC-ALZ consortia; Kehoe PG, Garcia-Ribas G, Sanchez-Juan P, Pastor P, Perez-Tur J, Pinol-Ripoll G, Lopez de Munain A, Garcia-Alberca JM, Bullido MJ, Alvarez V, Lleo A, Real LM, Mir P, Medina M, Scheltens P, Holstege H, Marquie M, Saez ME, Carracedo A, Amouyel P, Schellenberg GD, Williams J, Seshadri S, van Duijn CM, Mather KA, Sanchez-Valle R, Serrano-Rios M, Orellana A, Tarraga L, Blennow K, Huisman M, Andreassen OA, Posthuma D, Clarimon J, Boada M, van der Flier WM, Ramirez A, Lambert JC, van der Lee SJ, Ruiz A. Common variants in Alzheimer's disease and risk stratification by polygenic risk scores. Nat Commun. 2021 Jun 7;12(1):3417. doi: 10.1038/s41467-021-22491-8. PMID 34099642
- [Background] Jansen IE, van der Lee SJ, Gomez-Fonseca D, de Rojas I, Dalmasso MC, Grenier-Boley B, Zettergren A, Mishra A, Ali M, Andrade V, Bellenguez C, Kleineidam L, Kucukali F, Sung YJ, Tesi N, Vromen EM, Wightman DP, Alcolea D, Alegret M, Alvarez I, Amouyel P, Athanasiu L, Bahrami S, Bailly H, Belbin O, Bergh S, Bertram L, Biessels GJ, Blennow K, Blesa R, Boada M, Boland A, Buerger K, Carracedo A, Cervera-Carles L, Chene G, Claassen JAHR, Debette S, Deleuze JF, de Deyn PP, Diehl-Schmid J, Djurovic S, Dols-Icardo O, Dufouil C, Duron E, Duzel E; EADB consortium; Fladby T, Fortea J, Frolich L, Garcia-Gonzalez P, Garcia-Martinez M, Giegling I, Goldhardt O, Gobom J, Grimmer T, Haapasalo A, Hampel H, Hanon O, Hausner L, Heilmann-Heimbach S, Helisalmi S, Heneka MT, Hernandez I, Herukka SK, Holstege H, Jarholm J, Kern S, Knapskog AB, Koivisto AM, Kornhuber J, Kuulasmaa T, Lage C, Laske C, Leinonen V, Lewczuk P, Lleo A, de Munain AL, Lopez-Garcia S, Maier W, Marquie M, Mol MO, Montrreal L, Moreno F, Moreno-Grau S, Nicolas G, Nothen MM, Orellana A, Palhaugen L, Papma JM, Pasquier F, Perneczky R, Peters O, Pijnenburg YAL, Popp J, Posthuma D, Pozueta A, Priller J, Puerta R, Quintela I, Ramakers I, Rodriguez-Rodriguez E, Rujescu D, Saltvedt I, Sanchez-Juan P, Scheltens P, Scherbaum N, Schmid M, Schneider A, Selbaek G, Selnes P, Shadrin A, Skoog I, Soininen H, Tarraga L, Teipel S; GR@ACE study group; Tijms B, Tsolaki M, Van Broeckhoven C, Van Dongen J, van Swieten JC, Vandenberghe R, Vidal JS, Visser PJ, Vogelgsang J, Waern M, Wagner M, Wiltfang J, Wittens MMJ, Zetterberg H, Zulaica M, van Duijn CM, Bjerke M, Engelborghs S, Jessen F, Teunissen CE, Pastor P, Hiltunen M, Ingelsson M, Andreassen OA, Clarimon J, Sleegers K, Ruiz A, Ramirez A, Cruchaga C, Lambert JC, van der Flier W. Genome-wide meta-analysis for Alzheimer's disease cerebrospinal fluid biomarkers. Acta Neuropathol. 2022 Nov;144(5):821-842. doi: 10.1007/s00401-022-02454-z. Epub 2022 Sep 6. PMID 36066633
- [Background] Le Guen Y, Belloy ME, Grenier-Boley B, de Rojas I, Castillo-Morales A, Jansen I, Nicolas A, Bellenguez C, Dalmasso C, Kucukali F, Eger SJ, Rasmussen KL, Thomassen JQ, Deleuze JF, He Z, Napolioni V, Amouyel P, Jessen F, Kehoe PG, van Duijn C, Tsolaki M, Sanchez-Juan P, Sleegers K, Ingelsson M, Rossi G, Hiltunen M, Sims R, van der Flier WM, Ramirez A, Andreassen OA, Frikke-Schmidt R, Williams J, Ruiz A, Lambert JC, Greicius MD; Members of the EADB, GR@ACE, DEGESCO, DemGene, GERAD, and EADI Groups; Arosio B, Benussi L, Boland A, Borroni B, Caffarra P, Daian D, Daniele A, Debette S, Dufouil C, Duzel E, Galimberti D, Giedraitis V, Grimmer T, Graff C, Grunblatt E, Hanon O, Hausner L, Heilmann-Heimbach S, Holstege H, Hort J, Jurgen D, Kuulasmaa T, van der Lugt A, Masullo C, Mecocci P, Mehrabian S, de Mendonca A, Moebus S, Nacmias B, Nicolas G, Olaso R, Papenberg G, Parnetti L, Pasquier F, Peters O, Pijnenburg YAL, Popp J, Rainero I, Ramakers I, Riedel-Heller S, Scarmeas N, Scheltens P, Scherbaum N, Schneider A, Seripa D, Soininen H, Solfrizzi V, Spalletta G, Squassina A, van Swieten J, Tegos TJ, Tremolizzo L, Verhey F, Vyhnalek M, Wiltfang J, Boada M, Garcia-Gonzalez P, Puerta R, Real LM, Alvarez V, Bullido MJ, Clarimon J, Garcia-Alberca JM, Mir P, Moreno F, Pastor P, Pinol-Ripoll G, Molina-Porcel L, Perez-Tur J, Rodriguez-Rodriguez E, Royo JL, Sanchez-Valle R, Dichgans M, Rujescu D. Association of Rare APOE Missense Variants V236E and R251G With Risk of Alzheimer Disease. JAMA Neurol. 2022 Jul 1;79(7):652-663. doi: 10.1001/jamaneurol.2022.1166. PMID 35639372
- [Background] Bellenguez C, Kucukali F, Jansen IE, Kleineidam L, Moreno-Grau S, Amin N, Naj AC, Campos-Martin R, Grenier-Boley B, Andrade V, Holmans PA, Boland A, Damotte V, van der Lee SJ, Costa MR, Kuulasmaa T, Yang Q, de Rojas I, Bis JC, Yaqub A, Prokic I, Chapuis J, Ahmad S, Giedraitis V, Aarsland D, Garcia-Gonzalez P, Abdelnour C, Alarcon-Martin E, Alcolea D, Alegret M, Alvarez I, Alvarez V, Armstrong NJ, Tsolaki A, Antunez C, Appollonio I, Arcaro M, Archetti S, Pastor AA, Arosio B, Athanasiu L, Bailly H, Banaj N, Baquero M, Barral S, Beiser A, Pastor AB, Below JE, Benchek P, Benussi L, Berr C, Besse C, Bessi V, Binetti G, Bizarro A, Blesa R, Boada M, Boerwinkle E, Borroni B, Boschi S, Bossu P, Brathen G, Bressler J, Bresner C, Brodaty H, Brookes KJ, Brusco LI, Buiza-Rueda D, Burger K, Burholt V, Bush WS, Calero M, Cantwell LB, Chene G, Chung J, Cuccaro ML, Carracedo A, Cecchetti R, Cervera-Carles L, Charbonnier C, Chen HH, Chillotti C, Ciccone S, Claassen JAHR, Clark C, Conti E, Corma-Gomez A, Costantini E, Custodero C, Daian D, Dalmasso MC, Daniele A, Dardiotis E, Dartigues JF, de Deyn PP, de Paiva Lopes K, de Witte LD, Debette S, Deckert J, Del Ser T, Denning N, DeStefano A, Dichgans M, Diehl-Schmid J, Diez-Fairen M, Rossi PD, Djurovic S, Duron E, Duzel E, Dufouil C, Eiriksdottir G, Engelborghs S, Escott-Price V, Espinosa A, Ewers M, Faber KM, Fabrizio T, Nielsen SF, Fardo DW, Farotti L, Fenoglio C, Fernandez-Fuertes M, Ferrari R, Ferreira CB, Ferri E, Fin B, Fischer P, Fladby T, Fliessbach K, Fongang B, Fornage M, Fortea J, Foroud TM, Fostinelli S, Fox NC, Franco-Macias E, Bullido MJ, Frank-Garcia A, Froelich L, Fulton-Howard B, Galimberti D, Garcia-Alberca JM, Garcia-Gonzalez P, Garcia-Madrona S, Garcia-Ribas G, Ghidoni R, Giegling I, Giorgio G, Goate AM, Goldhardt O, Gomez-Fonseca D, Gonzalez-Perez A, Graff C, Grande G, Green E, Grimmer T, Grunblatt E, Grunin M, Gudnason V, Guetta-Baranes T, Haapasalo A, Hadjigeorgiou G, Haines JL, Hamilton-Nelson KL, Hampel H, Hanon O, Hardy J, Hartmann AM, Hausner L, Harwood J, Heilmann-Heimbach S, Helisalmi S, Heneka MT, Hernandez I, Herrmann MJ, Hoffmann P, Holmes C, Holstege H, Vilas RH, Hulsman M, Humphrey J, Biessels GJ, Jian X, Johansson C, Jun GR, Kastumata Y, Kauwe J, Kehoe PG, Kilander L, Stahlbom AK, Kivipelto M, Koivisto A, Kornhuber J, Kosmidis MH, Kukull WA, Kuksa PP, Kunkle BW, Kuzma AB, Lage C, Laukka EJ, Launer L, Lauria A, Lee CY, Lehtisalo J, Lerch O, Lleo A, Longstreth W Jr, Lopez O, de Munain AL, Love S, Lowemark M, Luckcuck L, Lunetta KL, Ma Y, Macias J, MacLeod CA, Maier W, Mangialasche F, Spallazzi M, Marquie M, Marshall R, Martin ER, Montes AM, Rodriguez CM, Masullo C, Mayeux R, Mead S, Mecocci P, Medina M, Meggy A, Mehrabian S, Mendoza S, Menendez-Gonzalez M, Mir P, Moebus S, Mol M, Molina-Porcel L, Montrreal L, Morelli L, Moreno F, Morgan K, Mosley T, Nothen MM, Muchnik C, Mukherjee S, Nacmias B, Ngandu T, Nicolas G, Nordestgaard BG, Olaso R, Orellana A, Orsini M, Ortega G, Padovani A, Paolo C, Papenberg G, Parnetti L, Pasquier F, Pastor P, Peloso G, Perez-Cordon A, Perez-Tur J, Pericard P, Peters O, Pijnenburg YAL, Pineda JA, Pinol-Ripoll G, Pisanu C, Polak T, Popp J, Posthuma D, Priller J, Puerta R, Quenez O, Quintela I, Thomassen JQ, Rabano A, Rainero I, Rajabli F, Ramakers I, Real LM, Reinders MJT, Reitz C, Reyes-Dumeyer D, Ridge P, Riedel-Heller S, Riederer P, Roberto N, Rodriguez-Rodriguez E, Rongve A, Allende IR, Rosende-Roca M, Royo JL, Rubino E, Rujescu D, Saez ME, Sakka P, Saltvedt I, Sanabria A, Sanchez-Arjona MB, Sanchez-Garcia F, Juan PS, Sanchez-Valle R, Sando SB, Sarnowski C, Satizabal CL, Scamosci M, Scarmeas N, Scarpini E, Scheltens P, Scherbaum N, Scherer M, Schmid M, Schneider A, Schott JM, Selbaek G, Seripa D, Serrano M, Sha J, Shadrin AA, Skrobot O, Slifer S, Snijders GJL, Soininen H, Solfrizzi V, Solomon A, Song Y, Sorbi S, Sotolongo-Grau O, Spalletta G, Spottke A, Squassina A, Stordal E, Tartan JP, Tarraga L, Tesi N, Thalamuthu A, Thomas T, Tosto G, Traykov L, Tremolizzo L, Tybjaerg-Hansen A, Uitterlinden A, Ullgren A, Ulstein I, Valero S, Valladares O, Broeckhoven CV, Vance J, Vardarajan BN, van der Lugt A, Dongen JV, van Rooij J, van Swieten J, Vandenberghe R, Verhey F, Vidal JS, Vogelgsang J, Vyhnalek M, Wagner M, Wallon D, Wang LS, Wang R, Weinhold L, Wiltfang J, Windle G, Woods B, Yannakoulia M, Zare H, Zhao Y, Zhang X, Zhu C, Zulaica M; EADB; GR@ACE; DEGESCO; EADI; GERAD; Demgene; FinnGen; ADGC; CHARGE; Farrer LA, Psaty BM, Ghanbari M, Raj T, Sachdev P, Mather K, Jessen F, Ikram MA, de Mendonca A, Hort J, Tsolaki M, Pericak-Vance MA, Amouyel P, Williams J, Frikke-Schmidt R, Clarimon J, Deleuze JF, Rossi G, Seshadri S, Andreassen OA, Ingelsson M, Hiltunen M, Sleegers K, Schellenberg GD, van Duijn CM, Sims R, van der Flier WM, Ruiz A, Ramirez A, Lambert JC. New insights into the genetic etiology of Alzheimer's disease and related dementias. Nat Genet. 2022 Apr;54(4):412-436. doi: 10.1038/s41588-022-01024-z. Epub 2022 Apr 4. PMID 35379992
- [Background] Le Guen Y, Luo G, Ambati A, Damotte V, Jansen I, Yu E, Nicolas A, de Rojas I, Peixoto Leal T, Miyashita A, Bellenguez C, Lian MM, Parveen K, Morizono T, Park H, Grenier-Boley B, Naito T, Kucukali F, Talyansky SD, Yogeshwar SM, Sempere V, Satake W, Alvarez V, Arosio B, Belloy ME, Benussi L, Boland A, Borroni B, Bullido MJ, Caffarra P, Clarimon J, Daniele A, Darling D, Debette S, Deleuze JF, Dichgans M, Dufouil C, During E, Duzel E, Galimberti D, Garcia-Ribas G, Garcia-Alberca JM, Garcia-Gonzalez P, Giedraitis V, Goldhardt O, Graff C, Grunblatt E, Hanon O, Hausner L, Heilmann-Heimbach S, Holstege H, Hort J, Jung YJ, Jurgen D, Kern S, Kuulasmaa T, Lee KH, Lin L, Masullo C, Mecocci P, Mehrabian S, de Mendonca A, Boada M, Mir P, Moebus S, Moreno F, Nacmias B, Nicolas G, Niida S, Nordestgaard BG, Papenberg G, Papma J, Parnetti L, Pasquier F, Pastor P, Peters O, Pijnenburg YAL, Pinol-Ripoll G, Popp J, Porcel LM, Puerta R, Perez-Tur J, Rainero I, Ramakers I, Real LM, Riedel-Heller S, Rodriguez-Rodriguez E, Ross OA, Royo LJ, Rujescu D, Scarmeas N, Scheltens P, Scherbaum N, Schneider A, Seripa D, Skoog I, Solfrizzi V, Spalletta G, Squassina A, van Swieten J, Sanchez-Valle R, Tan EK, Tegos T, Teunissen C, Thomassen JQ, Tremolizzo L, Vyhnalek M, Verhey F, Waern M, Wiltfang J, Zhang J; EADB; GR@ACE study group; DEGESCO consortium; DemGene; EADI; GERAD; Asian Parkinson's Disease Genetics consortium; Zetterberg H, Blennow K, He Z, Williams J, Amouyel P, Jessen F, Kehoe PG, Andreassen OA, Van Duin C, Tsolaki M, Sanchez-Juan P, Frikke-Schmidt R, Sleegers K, Toda T, Zettergren A, Ingelsson M, Okada Y, Rossi G, Hiltunen M, Gim J, Ozaki K, Sims R, Foo JN, van der Flier W, Ikeuchi T, Ramirez A, Mata I, Ruiz A, Gan-Or Z, Lambert JC, Greicius MD, Mignot E. Multiancestry analysis of the HLA locus in Alzheimer's and Parkinson's diseases uncovers a shared adaptive immune response mediated by HLA-DRB1*04 subtypes. Proc Natl Acad Sci U S A. 2023 Sep 5;120(36):e2302720120. doi: 10.1073/pnas.2302720120. Epub 2023 Aug 29. PMID 37643212
- [Background] de Rojas I, Moreno-Grau S, Tesi N, Grenier-Boley B, Andrade V, Jansen IE, Pedersen NL, Stringa N, Zettergren A, Hernandez I, Montrreal L, Antunez C, Antonell A, Tankard RM, Bis JC, Sims R, Bellenguez C, Quintela I, Gonzalez-Perez A, Calero M, Franco-Macias E, Macias J, Blesa R, Cervera-Carles L, Menendez-Gonzalez M, Frank-Garcia A, Royo JL, Moreno F, Huerto Vilas R, Baquero M, Diez-Fairen M, Lage C, Garcia-Madrona S, Garcia-Gonzalez P, Alarcon-Martin E, Valero S, Sotolongo-Grau O, Ullgren A, Naj AC, Lemstra AW, Benaque A, Perez-Cordon A, Benussi A, Rabano A, Padovani A, Squassina A, de Mendonca A, Arias Pastor A, Kok AAL, Meggy A, Pastor AB, Espinosa A, Corma-Gomez A, Martin Montes A, Sanabria A, DeStefano AL, Schneider A, Haapasalo A, Kinhult Stahlbom A, Tybjaerg-Hansen A, Hartmann AM, Spottke A, Corbaton-Anchuelo A, Rongve A, Borroni B, Arosio B, Nacmias B, Nordestgaard BG, Kunkle BW, Charbonnier C, Abdelnour C, Masullo C, Martinez Rodriguez C, Munoz-Fernandez C, Dufouil C, Graff C, Ferreira CB, Chillotti C, Reynolds CA, Fenoglio C, Van Broeckhoven C, Clark C, Pisanu C, Satizabal CL, Holmes C, Buiza-Rueda D, Aarsland D, Rujescu D, Alcolea D, Galimberti D, Wallon D, Seripa D, Grunblatt E, Dardiotis E, Duzel E, Scarpini E, Conti E, Rubino E, Gelpi E, Rodriguez-Rodriguez E, Duron E, Boerwinkle E, Ferri E, Tagliavini F, Kucukali F, Pasquier F, Sanchez-Garcia F, Mangialasche F, Jessen F, Nicolas G, Selbaek G, Ortega G, Chene G, Hadjigeorgiou G, Rossi G, Spalletta G, Giaccone G, Grande G, Binetti G, Papenberg G, Hampel H, Bailly H, Zetterberg H, Soininen H, Karlsson IK, Alvarez I, Appollonio I, Giegling I, Skoog I, Saltvedt I, Rainero I, Rosas Allende I, Hort J, Diehl-Schmid J, Van Dongen J, Vidal JS, Lehtisalo J, Wiltfang J, Thomassen JQ, Kornhuber J, Haines JL, Vogelgsang J, Pineda JA, Fortea J, Popp J, Deckert J, Buerger K, Morgan K, Fliessbach K, Sleegers K, Molina-Porcel L, Kilander L, Weinhold L, Farrer LA, Wang LS, Kleineidam L, Farotti L, Parnetti L, Tremolizzo L, Hausner L, Benussi L, Froelich L, Ikram MA, Deniz-Naranjo MC, Tsolaki M, Rosende-Roca M, Lowenmark M, Hulsman M, Spallazzi M, Pericak-Vance MA, Esiri M, Bernal Sanchez-Arjona M, Dalmasso MC, Martinez-Larrad MT, Arcaro M, Nothen MM, Fernandez-Fuertes M, Dichgans M, Ingelsson M, Herrmann MJ, Scherer M, Vyhnalek M, Kosmidis MH, Yannakoulia M, Schmid M, Ewers M, Heneka MT, Wagner M, Scamosci M, Kivipelto M, Hiltunen M, Zulaica M, Alegret M, Fornage M, Roberto N, van Schoor NM, Seidu NM, Banaj N, Armstrong NJ, Scarmeas N, Scherbaum N, Goldhardt O, Hanon O, Peters O, Skrobot OA, Quenez O, Lerch O, Bossu P, Caffarra P, Dionigi Rossi P, Sakka P, Mecocci P, Hoffmann P, Holmans PA, Fischer P, Riederer P, Yang Q, Marshall R, Kalaria RN, Mayeux R, Vandenberghe R, Cecchetti R, Ghidoni R, Frikke-Schmidt R, Sorbi S, Hagg S, Engelborghs S, Helisalmi S, Botne Sando S, Kern S, Archetti S, Boschi S, Fostinelli S, Gil S, Mendoza S, Mead S, Ciccone S, Djurovic S, Heilmann-Heimbach S, Riedel-Heller S, Kuulasmaa T, Del Ser T, Lebouvier T, Polak T, Ngandu T, Grimmer T, Bessi V, Escott-Price V, Giedraitis V, Deramecourt V, Maier W, Jian X, Pijnenburg YAL; EADB contributors; GR@ACE study group; DEGESCO consortium; IGAP (ADGC, CHARGE, EADI, GERAD); PGC-ALZ consortia; Kehoe PG, Garcia-Ribas G, Sanchez-Juan P, Pastor P, Perez-Tur J, Pinol-Ripoll G, Lopez de Munain A, Garcia-Alberca JM, Bullido MJ, Alvarez V, Lleo A, Real LM, Mir P, Medina M, Scheltens P, Holstege H, Marquie M, Saez ME, Carracedo A, Amouyel P, Schellenberg GD, Williams J, Seshadri S, van Duijn CM, Mather KA, Sanchez-Valle R, Serrano-Rios M, Orellana A, Tarraga L, Blennow K, Huisman M, Andreassen OA, Posthuma D, Clarimon J, Boada M, van der Flier WM, Ramirez A, Lambert JC, van der Lee SJ, Ruiz A. Author Correction: Common variants in Alzheimer's disease and risk stratification by polygenic risk scores. Nat Commun. 2023 Feb 9;14(1):716. doi: 10.1038/s41467-023-36192-x. No abstract available. PMID 36759603
- [Background] European Alzheimer's & Dementia Biobank Mendelian Randomization (EADB-MR) Collaboration; Luo J, Thomassen JQ, Bellenguez C, Grenier-Boley B, de Rojas I, Castillo A, Parveen K, Kucukali F, Nicolas A, Peters O, Schneider A, Dichgans M, Rujescu D, Scherbaum N, Jurgen D, Riedel-Heller S, Hausner L, Porcel LM, Duzel E, Grimmer T, Wiltfang J, Heilmann-Heimbach S, Moebus S, Tegos T, Scarmeas N, Clarimon J, Moreno F, Perez-Tur J, Bullido MJ, Pastor P, Sanchez-Valle R, Alvarez V, Boada M, Garcia-Gonzalez P, Puerta R, Mir P, Real LM, Pinol-Ripoll G, Garcia-Alberca JM, Royo JL, Rodriguez-Rodriguez E, Soininen H, Kuulasmaa T, de Mendonca A, Mehrabian S, Hort J, Vyhnalek M, van der Lee S, Graff C, Papenberg G, Giedraitis V, Boland A, Bacq-Daian D, Deleuze JF, Nicolas G, Dufouil C, Pasquier F, Hanon O, Debette S, Grunblatt E, Popp J, Benussi L, Galimberti D, Arosio B, Mecocci P, Solfrizzi V, Parnetti L, Squassina A, Tremolizzo L, Borroni B, Nacmias B, Sorbi S, Caffarra P, Seripa D, Rainero I, Daniele A, Masullo C, Spalletta G, Williams J, Amouyel P, Jessen F, Kehoe P, Tsolaki M, Rossi G, Sanchez-Juan P, Sleegers K, Ingelsson M, Andreassen OA, Hiltunen M, Van Duijn C, Sims R, van der Flier W, Ruiz A, Ramirez A, Lambert JC, Frikke-Schmidt R. Genetic Associations Between Modifiable Risk Factors and Alzheimer Disease. JAMA Netw Open. 2023 May 1;6(5):e2313734. doi: 10.1001/jamanetworkopen.2023.13734. PMID 37195665
- [Background] Lehmann S, Schraen-Maschke S, Vidal JS, Delaby C, Blanc F, Paquet C, Allinquant B, Bombois S, Gabelle A, Hanon O; The BALTAZAR Study Group. Head-to-Head Comparison of Two Plasma Phospho-tau Assays in Predicting Conversion of Mild Cognitive Impairment to Dementia. Clin Chem. 2023 Sep 1;69(9):1072-1083. doi: 10.1093/clinchem/hvad103. PMID 37654065
- [Background] Lehmann S, Schraen-Maschke S, Vidal JS, Delaby C, Blanc F, Paquet C, Allinquant B, Bombois S, Gabelle A, Hanon O. Plasma phosphorylated tau 181 predicts amyloid status and conversion to dementia stage dependent on renal function. J Neurol Neurosurg Psychiatry. 2023 Jun;94(6):411-419. doi: 10.1136/jnnp-2022-330540. Epub 2023 Apr 3. PMID 37012068
- [Background] Lehmann S, Schraen-Maschke S, Vidal JS, Allinquant B, Bombois S, Gabelle A, Hanon O. Plasma Abeta42/Abeta40 ratio is independent of renal function. Alzheimers Dement. 2023 Jun;19(6):2737-2739. doi: 10.1002/alz.12949. Epub 2023 Feb 12. No abstract available. PMID 36774628
- [Background] Lehmann S, Schraen-Maschke S, Vidal JS, Blanc F, Paquet C, Allinquant B, Bombois S, Gabelle A, Delaby C, Hanon O; BALTAZAR Study Group. Blood Neurofilament Levels Predict Cognitive Decline across the Alzheimer's Disease Continuum. Int J Mol Sci. 2023 Dec 11;24(24):17361. doi: 10.3390/ijms242417361. PMID 38139190
- [Derived] Duron E, Vidal JS, Grousselle D, Gabelle A, Lehmann S, Pasquier F, Bombois S, Buee L, Allinquant B, Schraen-Maschke S, Baret C, Rigaud AS, Hanon O, Epelbaum J. Somatostatin and Neuropeptide Y in Cerebrospinal Fluid: Correlations With Amyloid Peptides Abeta1-42 and Tau Proteins in Elderly Patients With Mild Cognitive Impairment. Front Aging Neurosci. 2018 Oct 1;10:297. doi: 10.3389/fnagi.2018.00297. eCollection 2018. PMID 30327597